CLINICAL TRIAL: NCT03153241
Title: Value of Subglottic Secretion Culture in Predicting Microbial Flora of Tracheal Secretions in Intubated Patients. a Prospective Observational Study
Brief Title: Subglottic Secretion Culture in Predicting Tracheal Microbial Flora
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, DE PASCALE GENNARO, Dr Giuseppe Bello (Principal-Investigator), Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 001
Record Dates: First submitted 2017-04-29; First posted 2017-05-15 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2019-07

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — subglottic secretions and tracheal aspirates
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Ventilator-associated pneumonia (VAP) continues to be a major cause of morbidity and mortality in the intensive care unit (ICU). Microaspiration of subglottic secretions accumulated above the endotracheal tube cuff is the primary route of bacterial entry into the lower respiratory tract.Therefore, removal of secretions from the subglottic spacehas been recommended as a preventive strategy to avoid microaspiration and VAP. In this context, whereas considerable literature exists on the use subglottic secretion drainage (SSD) in patients at risk for developing VAP, there is a lack of data on the bacterial growth in the subglottic fluid above the cuff.

The primary objective of the study will be to assess the value of subglottic secretion culture in predicting microbial flora of endotracheal aspirate samplein patients admitted to our ICU and under invasive mechanical ventilation for at least 48 hours. Secondary end-point will be to estimate the predictive value of subglottic secretion culture in identifying bacterial pathogens in the sub-population of patients who will develop VAP.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Invasive mechanical ventilation for at least 48 hours

Exclusion Criteria:

* age <18 years
* absence of informed consent
* pregnancy
* documented treatment-limitation orders in the patient's chart

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients under invasive mechanica ventilations for at least 48 hours
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-10-20 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Number of patients with the same pathogens in both subglottic secretions and endotracheal aspirates | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazioen Policlinico Universitario A. Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be made available to researchers upon a reasonable request

REFERENCES:
- [Derived] Bello G, Bisanti A, Giammatteo V, Montini L, Eleuteri D, Fiori B, La Sorda M, Spanu T, Grieco DL, Pennisi MA, De Pascale G, Antonelli M. Microbiologic surveillance through subglottic secretion cultures during invasive mechanical ventilation: a prospective observational study. J Crit Care. 2020 Oct;59:42-48. doi: 10.1016/j.jcrc.2020.05.013. Epub 2020 May 26. PMID 32516641